CLINICAL TRIAL: NCT00924222
Title: Organ Protection With Sevoflurane Postconditioning After Cardiac Surgery With Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFA-5-2007
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Cardiac On-pump Surgery
MeSH Terms: interventions — Sevoflurane; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Experimental)
  Interventions: Drug: Sevoflurane; Drug: Propofol
- Propofol (Experimental)
  Interventions: Drug: Sevoflurane; Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — Sedation with sevoflurane
Drug: Propofol — Sedation on intensive care unit with propofol

SUMMARY:
Organ protection, volatile anesthetics, postconditioning.

Sedation of patients on ICU after cardiac surgery with cardiopulmonary bypass with either propofol or sevoflurane. Evaluation of organ function and inflammatory mediators in the blood.

ELIGIBILITY:
Inclusion criteria:

* CABG and/or heart valve surgery with CPB
* Ejection fraction (EF) = 30%
* Canadian Cardiovascular Society (CCS) classification = 3
* Ages 18 to 90 years old

Exclusion criteria:

* Pulmonary disease: forced expiratory volume in one second (FEV1) < 80%; FEV1/forced vital capacity (FVC) < 70%
* Renal disease and/ or creatinine-clearance < 60 ml/min
* Previous cardiac surgery
* Emergency procedures
* Postoperative intra aortic balloon pump (IABP) requirement
* Myocardial infarction < 7d
* Steroid treatment
* Insulin-dependent diabetes
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-10; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Myocardial injury markers (myoglobin, creatine kinase, myocard specific creatine kinase, and troponin T) | Start and end of ICU stay

SECONDARY OUTCOMES:
Oxygenation index, postoperative pulmonary complications, ICU stay (days), length of hospitalisation | Start with surgery until end of hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland

REFERENCES:
- [Derived] Steurer MP, Steurer MA, Baulig W, Piegeler T, Schlapfer M, Spahn DR, Falk V, Dreessen P, Theusinger OM, Schmid ER, Schwartz D, Neff TA, Beck-Schimmer B. Late pharmacologic conditioning with volatile anesthetics after cardiac surgery. Crit Care. 2012 Oct 14;16(5):R191. doi: 10.1186/cc11676. PMID 23062276